CLINICAL TRIAL: NCT06249308
Title: A Multi-center, Perspective, Observational Case-control Study to Develop and Validate an Ovarian Cancer Early Detection Model Based on Peripheral Blood Multi-omic Analysis and Machine Learning
Brief Title: Liquid Biopsy-based Early Detection of Ovarian Cancer: a Proof-of-concept Study ( PROFOUND-OC )
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Shanghai Weihe Medical Laboratory Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hao Wen, Principal Investigator, Fudan University
Other Study IDs: PROFOUND -OC
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ovarian cancer: Participants with new diagnosis of ovarian cancer, from whom a peripheral blood sample will be collected.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood sample will be collected

SUMMARY:
This study is a multi-center, observational study aiming at developing a machine learning-based early detection model using prospectively collected liquid biopsy samples from newly diagnosed ovarian cancer.

DETAILED DESCRIPTION:
Peripheral blood samples from ovarian cancer (OC) patients will be prospectively collected to identify cancer-specific circulating signals by analyzing cell free DNA. Based on the comprehensive molecular profiling, a machine learning-driven noninvasive test will be trained and validated through a two-stage approach in clinically annotated individuals. Approximately 168 stage I-II OC patients will be enrolled in this study. Age-matched female controls included in model development were recruited in another study, which are volunteers without a cancer diagnosis after routine medical screening.

ELIGIBILITY:
Inclusion Criteria:

* 40-75 years old
* Clinically and/or pathologically diagnosed ovarian cancer
* No prior or undergoing any systemic or local antitumor therapy, including but not limited to surgical resection, radiochemotherapy, endocrinotherapy, targeted therapy, immunotherapy, interventional therapy, etc.
* Able to provide a written informed consent and willing to comply with all part of the protocol procedures

Exclusion Criteria:

* Pregnancy or lactating women
* Known prior or current diagnosis of other types of malignancies comorbidities
* Severe acute infection (e.g. severe or critical COVID-19, sepsis, etc.) or febrile illness (body temperature of ≥ 38.0 °C) within 14 days prior to blood draw
* Recipients of organ transplant or prior bone marrow transplant or stem cell transplant
* Recipients of blood transfusion within 30 days prior to study blood draw
* Recipients of therapy in past 14 days prior to blood draw, including oral or IV antibiotics, glucocorticoid, azacitidine, decitabine, procainamine, hydrazine, arsenic trioxide
* Other conditions that the investigators considered are not suitable for the enrollment

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed ovarian cancer or individuals with a high suspicion for OC will be invited to participate in this proof-of-concept study
Sampling Method: Non-Probability Sample
Enrollment: 168 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The performance of cfDNA methylation-based model for discriminating ovarian cancer versus non-cancer. | 12 months
  Sensitivities of cfDNA methylation-based model in detecting OC at specificity of 99% and 95%, respectively.

SECONDARY OUTCOMES:
The performance of model using multi-omics data for discriminating ovarian cancer versus non-cancer | 12 months
  Sensitivities of multi-omics model which combines methylation signature and fragmentomic features in detecting OC at specificity of 99% and 95%, respectively.
The performance of pre-defined model in clinical sub-groups of interest | 12 months
  Sensitivity of pre-defined model in different pathological subtypes or different age groups or tumor marker-negative cases.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Wen, M.D., Ph.D., Principal Investigator — Fudan University
Locations (3):
- China (3):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No